CLINICAL TRIAL: NCT02036255
Title: Prevention of Tunneled Cuffed Catheter Malfunction With Prophylactic Use of a Taurolidine Locking Solution Containing Urokinase : a Multicentric Randomized Controlled Trial
Brief Title: Prevention of Dialysis Catheter Malfunction With Prophylactic Use of a Taurolidine Containing Urokinase
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Bonkain Florence, Bonkain Florence, MD, UZ Brussel, Universitair Ziekenhuis Brussel
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TL-001
Record Dates: First submitted 2014-01-11; First posted 2014-01-14 (Estimated); Last update posted 2018-05-03 (Actual); Status verified 2018-05

CONDITIONS: Patency; Infection
Keywords: Prevention, Thrombosis, Hemodialysis, Vascular access device
MeSH Terms: conditions — Infections; Thrombosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Taurolidine Urokinase (Experimental): Taurolock Urokinase is used weekly in this arm substituting the classic Taurolock HEP500
  Interventions: Drug: Taurolidine Urokinase; Drug: Taurolidine Heparin
- Taurolidine Heparin (Active Comparator): Taurolock HEP 500 is used as locking solution after each dialysis session
  Interventions: Drug: Taurolidine Heparin

INTERVENTIONS:
Drug: Taurolidine Urokinase
  Other Names: Taurolock Urokinase 25,000
  Arms: Taurolidine Urokinase
Drug: Taurolidine Heparin
  Other Names: Taurolock HEP 500

SUMMARY:
The objective of our study is to investigate whether the substitution of the standard locking solution with a locking solution containing taurolidine and urokinase weekly (Taurolock ™ U 25,000 - www.taurolock.com ) reduces the rate of catheter dysfunction in hemodialysis patients with a history of TCC dysfunction requiring urokinase therapy.

ELIGIBILITY:
Inclusion Criteria:

* Adult, prevalent hemodialysis patients
* Informed and consented
* Hemodialysis 3x/week via a tunneled cuffed catheter
* Urokinase administration at least two times during the previous 6 months (with more than a week between 2 administrations)
* Adequate catheter function during the week before inclusion (defined by blood flow more than 250ml/min on each dialysis session and blood flow within 15% of the maximal blood flow after the last Urokinase administration)

Exclusion Criteria:

* Presence of heparin-induced thrombocytopenia
* Major hemorrhage or intracranial bleeding in the previous 3 months
* Pericarditis
* Intolerance to Taurolidine, citrate or to Urokinase
* Active catheter-related infection
* Catheter in the femoral vein

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2015-05; Primary Completion 2017-07 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Requirement of Urokinase | 6 months
  Requirement of Urokinase for thrombotic malfunction of dialyse catheter

SECONDARY OUTCOMES:
Removal of dialysis catheter | 6 months
  Removal of dialysis catheter for thrombosis and for bacteremia

OTHER OUTCOMES:
Comparison of the monthly cost of both procedures | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Florence FB Bonkain, MD, Principal Investigator — Universitair Ziekenhuis Brussel
Locations (9):
- Belgium (9):
  - Bracops Hospital, Anderlecht, Brussels Capital
  - Ixelles Hospital, Ixelles-Elsene, Brussels Capital
  - Brugman Hospital, Jette, Brussels Capital
  - Universitair Ziekenhuis Brussel, Jette, Brussels Capital
  - CHU Charleroi, Charleroi, Hainaut
  - CHWAPI, Tournai, Hainaut
  - UZ Antwerpen, Antwerp
  - Ixelles Hospital, Brussels
  - Ghent Hospital, Ghent

REFERENCES:
- [Background] Hemmelgarn BR, Moist LM, Lok CE, Tonelli M, Manns BJ, Holden RM, LeBlanc M, Faris P, Barre P, Zhang J, Scott-Douglas N; Prevention of Dialysis Catheter Lumen Occlusion with rt-PA versus Heparin Study Group. Prevention of dialysis catheter malfunction with recombinant tissue plasminogen activator. N Engl J Med. 2011 Jan 27;364(4):303-12. doi: 10.1056/NEJMoa1011376. PMID 21268722
- [Background] Trerotola SO, Johnson MS, Harris VJ, Shah H, Ambrosius WT, McKusky MA, Kraus MA. Outcome of tunneled hemodialysis catheters placed via the right internal jugular vein by interventional radiologists. Radiology. 1997 May;203(2):489-95. doi: 10.1148/radiology.203.2.9114110.
- [Background] Di Iorio BR, Bellizzi V, Cillo N, Cirillo M, Avella F, Andreucci VE, De Santo NG. Vascular access for hemodialysis: the impact on morbidity and mortality. J Nephrol. 2004 Jan-Feb;17(1):19-25. PMID 15151255
- [Derived] Bonkain F, Stolear JC, Catalano C, Vandervelde D, Treille S, Couttenye MM, Dhondt A, Libertalis M, Allamani M, Madhoun P, Van Craenenbroeck AH, Vanommeslaeghe F, Van Hulle F, Durieux P, Van Limberghen I, Tielemans C, Wissing KM. Prevention of tunneled cuffed catheter dysfunction with prophylactic use of a taurolidine urokinase lock: A randomized double-blind trial. PLoS One. 2021 May 20;16(5):e0251793. doi: 10.1371/journal.pone.0251793. eCollection 2021. PMID 34015014
- [Derived] Bonkain F, Van Hulle F, Janssens P, Catalano C, Allamani M, Stolear JC, Vandervelde D, Libertalis M, Treille S, Couttenye MM, Dhondt A, Van Biesen W, Fils JF, Tielemans C, Wissing KM. Urokinase-containing locking solution in the prevention of dialysis catheter dysfunction: a double blind randomized controlled trial. J Vasc Access. 2017 Sep 11;18(5):436-442. doi: 10.5301/jva.5000737. Epub 2017 Jun 14. PMID 28623638